CLINICAL TRIAL: NCT02850744
Title: Open-label, Non-randomized, Two-stage Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamic Effects of PQR309 in Patients With Progressive Glioblastoma
Brief Title: Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamic Effects of PQR309 in Glioblastoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: PIQUR Therapeutics AG (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQR309-004
Record Dates: First submitted 2016-03-24; First posted 2016-08-01 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm (Other): Open label, single arm including patients with progressive glioblastoma during or after temozolomide chemotherapy obtaining PQR309 80mg capsules.
  Interventions: Drug: PQR309

INTERVENTIONS:
Drug: PQR309 — 80mg capsules p.o. once daily and possibly Standard Treatment with temozolomide
  Other Names: temozolomide

SUMMARY:
PQR309 is an oral, dual pan-PI3K (phosphatidylinositol 3-kinase phosphoinositide 3-kinase) and mTOR (mammilian target of rapamycin) inhibitor that penetrates the blood-brain barrier at pharmacodynamically active concentrations. This study plans to evaluate PQR309 in treatment of patients with first progression of glioblastoma.

DETAILED DESCRIPTION:
Open-label, non-randomized, two-stage, multi-center study evaluating clinical efficacy, safety, pharmacokinetics and pharmacodynamic effects of PQR309 in patients with progressive glioblastoma during or after standard temozolomide chemoradiotherapy.

The first stage of the study will enroll a minimum of 18 patients with glioblastoma at first progression during or after temozolomide chemoradiotherapy or temozolomide only. Following the completion of recruitment of patients in the first stage of the study, the decision will be made by the study team (study investigators and the sponsor), based on the continuous evaluation of safety and efficacy data, whether to continue recruitment of patients in the second stage while awaiting the data analyses. 17 additional patients may be enrolled for the second stage of the study, for a minimum of 35 patients in total. All patients evaluable for the primary endpoint will be followed until disease progression or death.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed glioblastoma at first progression following or during standard temozolomide chemoradiotherapy (TMZ/RTTMZ)
2. older than 18 years of age
3. Radiographic demonstration of disease progression by RANO criteria
4. Only for patients of the surgical cohort:

   * Eligible for open resection of progressive tumor according to standard practice of the study center
   * Availability of adequate surgical tissue sample for the evaluation of concentration of PQR309 in the tumor and its PD effect
   * Patients treated with PQR309 after incomplete surgical resection may still have measurable disease according to RANO criteria and may therefore be evaluable for evaluation of response to treatment with PQR309 according to RANO criteria. The best response in patients treated with PQR309 after complete surgical resection is stable disease. All patients can be assessed for PFS6.
5. Only for patients of the non-surgical cohort:

   - Presence of at least one lesion of bi-dimensionally measurable disease by MRI with a contrast-enhancing tumor of at least 1 cm (10 mm) in the longest diameter on baseline MRI is required for patients who do not undergo surgery at relapse. For patients who undergo surgery for recurrence but do not participate in the presurgical PQR309 dosing cohort, the same rules regarding response assessment as in the surgical cohort apply. All patients can be assessed for PFS6.
6. Patient must have at least 1 formalin-fixed paraffin-embedded archival tumor tissue block representative of glioblastoma available from the first surgical resection of glioblastoma.
7. One prior systemic therapy regimen: patients must have received at least one dose of TMZ in the first line therapy. More than 6 cycles and alternative dosing regiments of TMZ are allowed.
8. If receiving corticosteroids, patients must have been on a stable or decreasing dose of corticosteroids and no more than 8 mg dexamethasone equivalent for ≥ 5 days prior to baseline MRI.
9. Karnofsky Performance Score (KPS) >70%.
10. More than 12 weeks from radiotherapy (RT)
11. More than 4 weeks from last administration of TMZ
12. More than 4 weeks from any investigational agent (at the judgment of the investigator and in agreement with lead investigator and PIQUR)
13. Adequate hematological, liver and renal function defined as follows:

    Absolute neutrophil count (ANC) ≥1.5x109/l, platelets ≥ 100x109/l, hemoglobin ≥ 100g/L. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN Serum Creatinine ≤ 1.5 times ULN
14. Able and willing to swallow and retain oral medication
15. Female and male patients of reproductive potential must agree to use effective contraception from screening until 90 days after discontinuing study treatment*
16. Willing and able to sign the informed consent and to comply with the protocol for the duration of the study

Exclusion Criteria:

1. Second or later glioblastoma relapse
2. Received more than one systemic treatment regimen for glioblastoma
3. Patients receiving enzyme-inducing anti-epileptic drug (EIAED) within 7 days of the first dose of PQR309
4. Patient is taking a drug with known risk to promote QT prolongation and Torsades de Pointes.
5. Patient is currently using herbal preparations or medications. Patient should stop using herbal medications 7 days prior to the first dose of the study drug
6. Patients with glioblastoma known to contain IDH1 or 2 mutation
7. Other concomitant anti-tumor therapy as determined by the study team
8. Prior treatment with intracerebral agents, e.g. prolifeprospan 20 with carmustine wafer
9. Patients unable to undergo contrast-enhanced MRI
10. Fasting glucose > 7.0 mmol/L or HbA1c > 6.4%.
11. Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders.
12. Anxiety ≥CTC AE grade 3
13. Patient has an uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, known HIV infection, chronic liver disease, chronic renal disease, pancreatitis, chronic pulmonary disease, active cardiac disease or cardiac dysfunction, interstitial lung disease, active autoimmune disease, uncontrolled diabetes, neuropsychiatric or social situations that would limit compliance with the study requirements
14. Presence of gastrointestinal disease or any other condition that could interfere significantly with the absorption of the study drug.
15. Concomitant treatment with medicinal products that increase the pH (reduce acidity) of the upper gastrointestinal tract, including, but not limited to, proton-pump inhibitors (e.g. omeprazole), H2-antagonists (e.g. ranitidine) and antacids. Patients may be enrolled in the study after a wash-out period sufficient to terminate their effect (See section 11.2.2.8).Women who are pregnant or breast feeding,
16. Women able to conceive and unwilling to practice an effective method of birth control* from screening until 90 days after discontinuing study treatment (women of childbearing potential** must have a negative urine or serum pregnancy test within 7 days prior to first dose of PQR309

    * Adequate contraception is defined as surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), or double-barrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap). Male patients must agree to use condoms as contraception method.

      * Child-bearing potential for the sake of this study is defined as sexually mature women who have not undergone a hysterectomy, have not been naturally postmenopausal for at least 12 consecutive months or have a serum FSH < 40 mIU/ml.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 6 months (PFS6) based on RANO criteria [30]glioblastoma, using progression-free survival rate at 6 months (PFS6) based on RANO criteria [30] | Change to base line of contrast MRI scans and incorporated clinical signs will be assessed on Day 1 of Cycle 1 and on Day 1 of every following cycle and at the end of treatment which can be up to 24 months after
  Non Surgical Cohort, Tumor response evaluation according to RANO criteria
Progression-free survival rate at 6 months (PFS6) based on RANO criteria [30]glioblastoma, using progression-free survival rate at 6 months (PFS6) based on RANO criteria [30] | Change to base line of contrast MRI scans and incorporated clinical signs will be assessed on Day1 pre-surgery, Day 4 post-surgery and 30 days after surgery and thereafter every 8 weeks (+/-7 days) until end of treatment up to 24mths
  Surgical Cohort, Tumor response evaluation according to RANO criteria

SECONDARY OUTCOMES:
Number of Adverse Events and Serious Adverse Events as related to the study medication | Cycle 1 on Day 1,2,8 and 15, on Cycle 2 and following cycles on Day 1 and 15 und 30 days after end of treatmen which can up to 24 months
  Non surgical cohort
Number of Adverse Events and Serious Adverse Events as related to the study medication | Assessment on Day 1,2 pre-surgery, Day3 surgery, Day4 post -surgery and 30 days after surgery, Cycle 2 on Day 1 and 15 and 30 days after end of treatment which can be up to 24 months
  Surgical cohort
Changes in pulse rate | Assessment on Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical Cohort
Changes in pulse rate | Assessment will during Cycle 1 on day 1,8,15, Cycle 2 day 1, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment and 30 days after last treatment
  Non-surgical cohort
Changes in blood pressure | Assessment on Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical cohort
Changes in blood pressure | Assessment will during Cycle 1 on day 1,8,15, Cycle 2 day 1, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment and 30 days after last treatment
  Non-surgical cohort
Changes in body weight | Assessment on Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical cohort
Changes in body weight | Assessment will during Cycle 1 on day 1,8,15, Cycle 2 day 1, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment and 30 days after last treatment
  Non-surgical cohort
Changes in temperature | Assessment on Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical Cohort
Changes in temperature | Assessment will during Cycle 1 on day 1,8,15, Cycle 2 day 1, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment and 30 days after last treatment
  Non-surgical cohort
Changes in ECG | Assessment on Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical Cohort
Changes in ECG | Assessment will during Cycle 1 on day 1,8,15, Cycle 2 day 1, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment and 30 days after last treatment
  Non-surgical cohort
Physical examination according to Karnofsky Performance Status | Assessment on Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical cohort
Physical examination according to Karnofsky Performance Status | Assessment will during Cycle 1 on day 1,8,15, Cycle 2 day 1, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment and 30 days after last treatment
  Non-surgical cohort
Depression Test (PHQ-9) | Assessment on Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical cohort
Depression test PHQ-9 | CAssessment will during Cycle 1 on day 1,8,15, Cycle 2 day 1, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment and 30 days after last treatment
  Non-surgical cohort
Generalized Anxiety Disorder mood scale score (GAD7) | Assessment on Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical Cohort
Generalized Anxiety Disorder mood scale score (GAD) | Cycle 1Assessment will during Cycle 1 on day 1,8,15, Cycle 2 day 1, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment and 30 days after last treatment
  Non-surgical cohort
Changes in routine blood chemistry | Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical cohort
Changes in routine blood chemistry | Cycle 1 on day 1,8,15, Cycle 2 day 1& 15, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment & 30 days after last treatment
  Non-surgical cohort
Changes in hematology | Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical cohort
Changes in hematology | Cycle 1 on day 1,8,15, Cycle 2 day 1& 15, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment & 30 days after last treatment
  Non-surgical cohort
Changes of urinalysis | Day1,2 pre-surgery, Day 3 surgery and Day 4 post-surgery and 30 days after surgery
  Surgical cohort
Changes of urinalysis | Cycle 1 on day 1,8,15, Cycle 2 day 1& 15, Cycle 3 und follow up cycles on day 1 up to 24 weeks, end of treatment & 30 days after last treatment
  Non-surgical cohort
Change of Insulin/Glucose/C-Peptide | Day 1: at pre-dose and 0.5, 1, 2, 4, 6, 8 hours post-dose (± 5 minutes) Day 2: at pre-dose (= 24 hour post first dose on Day 1) (± 5 minutes)& 3 - Pre-dose, and 1hr post dose. Day 4 - 24hr post last dose on Day 3
  Surgical cohort
Change of Insulin/Glucose/C-Peptide | Cycle 1 Day 1 - Pre-dose, 1hr post dose. Day 2 - 24hr post-dose. Cycle 2 Day 1 - pre-dose.
  Non- surgical cohort
Change of Haemostasis | Cycle 1 Day 1 - Pre-dose, 1hr post dose. Day 2 - 24hr post-dose. Cycle 2 Day 1 - pre-dose.
  Non- surgical cohort
Change of Haemostasis | Cycle 1 Day 1 - Pre-dose, 1hr post dose. Day 2 - 24hr post-dose. Cycle 2 Day 1 pre-dose.
  Surgical cohort
Determination of cmax | Day 1: at pre-dose ,0.5, 1, 2, 4, 6, 8 hours post-dose ;Day 2: at pre-dose (= 24 hour post first dose on Day 1);Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose; Day 4: at 24h after the last dose
  Surgical cohort
Determination of cmax | Day 1: at pre-dose and 0.5, 1, 2, 4, 6, 8 hours post-dose; Day 2: at pre-dose (= 24 hour post first dose on Day 1), Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose, Day 4: at 24h after the last dose
  Surgical cohort
Determination of AUC0-24 | Day 1: at pre-dose ,0.5, 1, 2, 4, 6, 8 hours post-dose ;Day 2: at pre-dose (= 24 hour post first dose on Day 1);Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose; Day 4: at 24h after the last dose
  Non-surgical cohort
Determination of AUC0-24 | Day 1: at pre-dose ,0.5, 1, 2, 4, 6, 8 hours post-dose ;Day 2: at pre-dose (= 24 hour post first dose on Day 1);Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose; Day 4: at 24h after the
  Non-surgical cohort
Determination of tmax | Day 1: at pre-dose ,0.5, 1, 2, 4, 6, 8 hours post-dose ;Day 2: at pre-dose (= 24 hour post first dose on Day 1);Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose; Day 4: at 24h after the
  Non-surgical cohort
Determination of AUClast | Day 1: at pre-dose ,0.5, 1, 2, 4, 6, 8 hours post-dose ;Day 2: at pre-dose (= 24 hour post first dose on Day 1);Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose; Day 4: at 24h after the
  Non-surgical cohort
Determination of tmax | Day 1: at pre-dose ,0.5, 1, 2, 4, 6, 8 hours post-dose ;Day 2: at pre-dose (= 24 hour post first dose on Day 1);Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose; Day 4: at 24h after the last dose
  Surgical cohort
Determination of AUClast | Day 1: at pre-dose and 0.5, 1, 2, 4, 6, 8 hours post-dose; Day 2: at pre-dose (= 24 hour post first dose on Day 1), Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose, Day 4: at 24h after the last dose
  Surgical cohort
Determination of AUC0-∞ | Day 1: at pre-dose ,0.5, 1, 2, 4, 6, 8 hours post-dose ;Day 2: at pre-dose (= 24 hour post first dose on Day 1);Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose; Day 4: at 24h after the last dose
  Surgical cohort
Determination of AUC0-∞ | Day 1: at pre-dose ,0.5, 1, 2, 4, 6, 8 hours post-dose ;Day 2: at pre-dose (= 24 hour post first dose on Day 1);Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose; Day 4: at 24h after the
  Non-surgical cohort
Determination of t½ | Day 1: at pre-dose ,0.5, 1, 2, 4, 6, 8 hours post-dose ;Day 2: at pre-dose (= 24 hour post first dose on Day 1);Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose; Day 4: at 24h after the last dose
  Surgical cohort
Determination of t½ | Day 1: at pre-dose ,0.5, 1, 2, 4, 6, 8 hours post-dose ;Day 2: at pre-dose (= 24 hour post first dose on Day 1);Day 3:at pre-dose, 0.5h, 1.0h, 2h, 4h, 6h, 8h post-dose; Day 4: at 24h after the
  Non-surgical cohort
Assessment of tumor concentration, | On day of surgery (day 3)
  Surgical cohort only
Assessment of PQR309 concentration in cerebrospinal fluid Day 3,pre-dose,0.5h, 1h, 2h, 4h, 6h, 8h post-dose Day 4 24h after the last dose given | On day of surgery (day 3)
  Surgical cohort only
Assessment of PQR309 Skin concentration | On day of surgery (day 3)
  Surgical cohort only
Overall Response Rate (ORR) including complete and partial Response based on RANO criteria | Change to base line of contrast MRI scans and incorporated clinical signs will be assessed on Day 1 of Cycle 1 and on Day 1 of every following cycle and at the end of treatment which can be up to 24 months after
  Surgical and Non-surgical Cohort
Duration of response (DOR) based on RANO criteria | of contrast MRI scans and incorporated clinical signs will be assessed on Day 1 of Cycle 1 and on Day 1 of every following cycle and at the end of treatment which can be up to 24 months after
  Surgical and non-surgical cohort
Progression-free survival at 3 months (PFS3) based on RANO criteria | of contrast MRI scans and incorporated clinical signs will be assessed on Day 1 of Cycle 1 and on Day 1 of every following cycle and at the end of treatment which can be up to 24 months after
  Surgical and non surgical cohort

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, Professor, Principal Investigator — University Hospital Zurich, Neurology
Locations (1):
- University Hospital Zurich, Neurology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No